CLINICAL TRIAL: NCT06148441
Title: Risk Factors and Novel Biomarkers Associated With In-stent Restenosis After Percutaneous Coronary Intervention
Brief Title: Role of Novel Biomarkers Associated With In-stent Restenosis After Percutaneous Coronary Intervention
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Elhussein Ahmed Mohamed, Doctor, Assiut University
Other Study IDs: novel biomarkers and ISR
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: In-stent Restenosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: bone morphogenetic protein-2 (BMP-2) — novel biomarkers associated with in-stent restenosis after percutaneous coronary intervention
  Other Names: novel biomarkers (high-sensitivity CRP (hs-CRP)

SUMMARY:
To study the relation between ISR and neutrophil-to-lymphocyte ratio (NLR), novel biomarkers (high-sensitivity CRP (hs-CRP), bone morphogenetic protein-2 (BMP-2) and other risk factors (age, sex, smoking, hypertension, diabetes, obesity, chronic kidney disease (CKD; creatinine clearance).

DETAILED DESCRIPTION:
Coronary artery disease (CAD) is the most common cardiovascular disease and remains a major global public health problem [1]. Due to the benefits of a shorter procedure time and reduced invasiveness, percutaneous coronary intervention (PCI) has become the predominant choice for coronary revascularization in patients with both stable and unstable CAD. However, in-stent restenosis (ISR) remains the leading problem after PCI, especially in patients with type 2 diabetes mellitus (T2DM) [2,3]. Diabetes mellitus is also regarded as one of the most powerful clinical predictors of ISR after drug-eluting stent (DES) implantation, which was also the case during the BMS era[4,5]. Although interventional approaches and pharmacological therapies have improved in recent years [6], ISR remains a problem; therefore, it is still important and useful to identify biomarkers that can predict ISR.

Bone morphogenetic protein-2 (BMP-2), a member of the transforming growth factor (TGF) superfamily, plays a significant role in both physiological and pathological vascular processes [7,8]. Recent studies have found that BMP-2 signalling is also associated with vascular disease, including atherosclerosis, vascular inflammation, vascular calcification and plaque instability [9,10]. Although diabetes has a well-known association with an increased risk for cardiovascular disease, the associated pathogenesis is not completely understood. In vitro studies have shown that high glucose concentrations are associated with increased expression of BMP-2 [11]. Plasma BMP-2 concentrations positively correlated with plaque burden and plaque calcification, which also positively correlated with plasma HbA1c. These findings suggest that BMP-2 may have a role in hyperglycaemia-induced calcification [12]. Endothelial dysfunction caused by stent implantation induces inflammation, which may also stimulate SMC proliferation [13-14]. Previous studies have revealed that chronic inflammation and fibrin deposition frequently persist for approximately 3 months after DES implantation, following the replacement of type III collagen by type I collagen and vascular smooth muscle cell (VSMC) proliferation [15]. Although the timing of intimal SMC proliferation is not clear, the migration of cells from within the plaque to the expanding neointima is the dominant factor that leads to ISR [15, 16]. BMP-2 is highly expressed in human vessels, and VSMCs are a significant source of BMP-2 [17,18]. In addition, several studies have indicated that BMP-2 promotes the migration of VSMCs by inducing the SMC phenotype towards a synthetic state and is closely associated with inflammation [8,19].Several studies have reported the clinical impact of hs-CRP levels in the chronic phase on clinical outcomes in CAD patients who underwent PCI. Hsieh et al. reported that higher hs-CRP levels (>3.0 mg/L) at 9-month follow-up angiography after PCI were associated with higher incidence of overall mortality and future clinical cardiovascular outcomes, including restenosis [20]. These findings indicate that hs-CRP could offer a useful biomarker for predicting the risk of adverse cardiovascular events or mortality in CAD patients after PCI.

These results are supported by the fact that inflammation underlies many of the processes contributing to atherogenesis and plaque destabilization. It has been indicated that hs-CRP may contribute to the development of arteriosclerosis in the presence of modified low-density lipoprotein (LDL) such as oxidized LDL [21].

This suggests that the type of stent is only one factor to consider when searching for additional promoters of ISR. The present study aimed to detect the clinical, biological, imagistic and procedural factors associated with ISR.

What is the meaning of ISR?ISR was defined as the narrowing of the lumen diameter of the target vessel ≥50%, including the coronary arteries in the stent and the ≤5 mm area adjacent to the stent [8]

ELIGIBILITY:
Inclusion Criteria:

* Patients with previously implanted 3rd generation DES (Sirolimus, Biolimus, Everolimus, Zotarolimus), whatever the duration since implantation or the setting of implantation or the number of implanted stents, and who are presenting to our institute along the coming two years for CA±PCI because of recurrent chest pain with suspicious of ISR or other newly developed lesions.

Exclusion Criteria:

* • Previous CABG

  * ACS within the last 2ms before the index CA for those undergoing assessment of hs-CRP & BMP-2
  * Heart failure with reduced EF<40%
  * Severe liver or kidney disease
  * Autoimmune, inflammatory, or malignant diseases
  * Non-available previous PCI CD & report

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with previously implanted 3rd generation DES (Sirolimus, Biolimus, Everolimus, Zotarolimus), whatever the duration since implantation or the setting of implantation or the number of implanted stents, and who are presenting to our institute along the coming two years for CA±PCI because of recurrent chest pain with suspicious of ISR or other newly developed lesions.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Role of novel biomarkers (high-sensitivity CRP (hs-CRP), bone morphogenetic protein-2 (BMP-2) associated with in-stent restenosis after percutaneous coronary intervention | Baseline
  Analysis of high-sensitivity CRP (hs-CRP), bone morphogenetic protein-2 (BMP-2) and incidence of ISR after percutaneous coronary intervention

REFERENCES:
- [Background] Assimes TL, Roberts R. Genetics: Implications for Prevention and Management of Coronary Artery Disease. J Am Coll Cardiol. 2016 Dec 27;68(25):2797-2818. doi: 10.1016/j.jacc.2016.10.039. PMID 28007143
- [Background] Mauri L, Silbaugh TS, Wolf RE, Zelevinsky K, Lovett A, Zhou Z, Resnic FS, Normand SL. Long-term clinical outcomes after drug-eluting and bare-metal stenting in Massachusetts. Circulation. 2008 Oct 28;118(18):1817-27. doi: 10.1161/CIRCULATIONAHA.108.781377. Epub 2008 Oct 13. PMID 18852368
- [Background] Kitoga M, Pasquet A, Preumont V, Kefer J, Hermans MP, Vanoverschelde JL, Buysschaert M. Coronary in-stent restenosis in diabetic patients after implantation of sirolimus or paclitaxel drug-eluting coronary stents. Diabetes Metab. 2008 Feb;34(1):62-7. doi: 10.1016/j.diabet.2007.09.002. PMID 18069029
- [Background] Csiszar A, Smith KE, Koller A, Kaley G, Edwards JG, Ungvari Z. Regulation of bone morphogenetic protein-2 expression in endothelial cells: role of nuclear factor-kappaB activation by tumor necrosis factor-alpha, H2O2, and high intravascular pressure. Circulation. 2005 May 10;111(18):2364-72. doi: 10.1161/01.CIR.0000164201.40634.1D. Epub 2005 Apr 25. PMID 15851600